CLINICAL TRIAL: NCT02969577
Title: Staying Strong and Healthy During Androgen Deprivation Therapy (ADT) for Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004205; R01NR014518 (NIH)
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: Androgen deprivation therapy; ADT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Resistance Training; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staying Strong & Healthy Intervention (SS&H) (Experimental): Participants will take part in a 6-month exercise program and diet and nutrition coaching program. Also part of this arm is a nutritional and lifestyle counseling program to be lead by a member of the study team. Participants will also receive the usual care they would normally receive if not taking part in this study.
  Interventions: Behavioral: Exercise Program; Behavioral: Diet and Nutrition Coaching; Other: Usual Care with Attention
- Usual Care with Attention (UCA) (Active Comparator): Participants will receive the usual care they would normally receive if not taking part in this study.
  Interventions: Other: Usual Care with Attention

INTERVENTIONS:
Behavioral: Exercise Program — Participants will have a personal training session at the first visit. A member of the study team will discuss strength training and cardiovascular workouts for them to complete over the first 6 months of the study. A member of the study team will then talk with the participant every week for the first 3 months and monthly afterwards until month 6. Participants will be sent exercise videos and be given recommendations for the exercise program via phone calls and will be tailored to the individual. Videos and recommendations will be sent directly to the participant's smartphone.
  Arms: Staying Strong & Healthy Intervention (SS&H)
Behavioral: Diet and Nutrition Coaching — Diet and nutrition coaching session with an overview of resources on the smartphone. Over the first 6 months, participants will receive healthy recipes and nutritional information on the smartphone.
  Arms: Staying Strong & Healthy Intervention (SS&H)
Other: Usual Care with Attention — Participants will receive the usual care for men undergoing ADT. This includes monitoring blood work and answering questions about how they are feeling. Participants will be directed to the IMPACT website for education materials on prostate cancer.

SUMMARY:
The purpose of this study is to learn if lifestyle changes and counseling along with standard medical care, compared to standard medical care alone, can prevent heart problems and diabetes in men who are receiving ADT for prostate cancer treatment.

DETAILED DESCRIPTION:
Prostate cancer is a very treatable cancer but those treatments can have long-lasting effects. A kind of hormone therapy called Androgen Deprivation Therapy (ADT) is often used along with other treatments like radiation and has been shown to improve survival. However, ADT can have negative effects especially on the heart and metabolism (the body's system for using and storing energy).

Participation in this study will last for up to 12 months. The study is looking at two different approaches to treating men who are undergoing ADT:

1. Staying Strong & Healthy Intervention + Usual Care
2. Usual Care

All participants will have blood drawn and be asked questions about how they are feeling during their participation. The men in the Staying Strong & Healthy Intervention group will also take part in a diet and exercise program and receive counseling from a member of the study team.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer
* Starting or have started ADT (oral or injection) for prostate cancer treatment within the last 3 months
* Re-initiating ADT after being on holiday for longer than their ADT dosage (e.g. If the man's dosage is every six months and he has been off ADT for more than six he is eligible);
* Able to speak and read in English or Spanish
* Reachable consistently by telephone
* Able to travel to KUMC

Exclusion Criteria:

* Not diagnosed with prostate cancer
* Not receiving or planning to receive ADT for prostate cancer treatment within the last three months
* Initiating ADT for prostate cancer prior to the previous 3 months or are not on ADT holiday
* Not able to speak and read in English or Spanish
* Not reachable consistently by telephone
* Not able to travel to the study site for data collection

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in LDL | Change from Baseline to Month 12

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Change from Baseline to Month 6
Change in Body Mass Index (BMI) | Change from Baseline to Month 12
Change in Lipid Profile | Change from Baseline to Month 6
Change in Lipid Profile | Change from Baseline to Month 12
Change in Waist/Hip Circumference | Change from Baseline to Month 6
Change in Waist/Hip Circumference | Change from Baseline to Month 12
Change in Glucose | Change from Baseline to Month 6
Change in Glucose | Change from Baseline to Month 12
Change in Health Related Quality | Change from Baseline to Month 6
  Quality of life will be measured using the SF-12 and Expanded Prostate Cancer Index Composite. The two are scored together and result in a composite score. Scores can range from 0-100. The higher the score the better the quality of life.
Change in Health Related Quality | Change from Baseline to Month 12
  Quality of life will be measured using the SF-12 and Expanded Prostate Cancer Index Composite. The two are scored together and result in a composite score. Scores can range from 0-100. The higher the score the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Maliski, PhD, RN, FAAN, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - University of Kansas Medical Center, Kansas City, Kansas